CLINICAL TRIAL: NCT05903274
Title: A Phase 1 Open-label, Dose-escalation, Safety, and Tolerability Study of JSP191 As a Second-line Therapy in Subjects with Lower-Risk Myelodysplastic Syndrome (LR-MDS)
Brief Title: JSP191 (briquilimab) in Subjects with LR-MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a lack of improvement in clinical efficacy outcomes.
Sponsor: Jasper Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JSP-CP-008
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Lower-risk Myelodysplastic Syndrome
Keywords: LR-MDS; cytopenia
MeSH Terms: conditions — Cytopenia

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation/de-escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- JSP191 (Experimental): This study will explore up to 5 ascending dose levels (Cohorts 1, 2, 3, 4, and 5) and subjects will receive JSP191 on Day 1 on each 8-week cycle for 4 consecutive cycles.
  Interventions: Drug: JSP191

INTERVENTIONS:
Drug: JSP191 — Subjects will receive intravenous JSP191
  Other Names: JSP191 (Briquilimab)

SUMMARY:
A Phase 1 study in subjects with LR-MDS to assess the safety and tolerability of JSP191 as a second-line therapy.

DETAILED DESCRIPTION:
An open-label, single-arm, dose-escalation study designed to determine the potential safety, efficacy, maximum tolerated dose (MTD) or optimal biologic dose (OBD), and recommended phase 2 dose (RP2D) of JSP191 (briquilimab) monotherapy for LR-MDS subjects with documented cytopenia (red blood cell-transfusion dependent, thrombocytopenia, and/or neutropenia).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* MDS with IPSS-R very low, low, or intermediate risk features
* Symptomatic cytopenias
* Women of childbearing potential (WOCBP) must agree to use an oral or implanted contraceptive, a double-barrier method of birth control, or an intrauterine device upon enrollment and through 3 months after receiving the last dose of JSP191
* Women not of childbearing potential must be post-menopausal (no menstrual period for a minimum of 12 months) or surgically sterilized and have a negative serum pregnancy test upon study entry
* Male subjects must be surgically sterile or willing to use contraception upon enrollment and through 3 months after receiving the last dose of JSP191
* Must be willing and able to provide informed consent

Exclusion Criteria:

* Anemia secondary to iron deficiency, vitamin B12 deficiency, or folate deficiency
* Prior allogeneic or autologous stem cell transplant
* Known history of human immunodeficiency virus (HIV) (no laboratory testing is required), or active infection with hepatitis B or hepatitis C
* Pregnant women or women who are nursing and do not wish to discontinue breastfeeding
* Any other medical condition that, in the opinion of the Investigator, could pose a significant safety risk to the subject or jeopardize the integrity of the study
* Subjects who, in the opinion of the Investigator, may not be able to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of JSP191 | 32 weeks
  Assessed by the frequency, duration, and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Jasper Therapeutics
Locations (2):
- United States (2):
  - Memorial Healthcare System, Hollywood, Florida
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.jaspertherapeutics.com/